CLINICAL TRIAL: NCT01582581
Title: Information Technology Enabled Treatment of Adolescent Depression
Brief Title: Study of Technology-assisted Treatment of Adolescent Depression
Acronym: iTAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iHope Network, Inc. (Industry)
Collaborators: Woburn Pediatric Associates (Unknown); UConn Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VHS 85350-02
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Major Depressive Disorder
Keywords: mental health; depression; behavioral health; cognitive behavioral therapy; CBT; computer-assisted psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major; Psychological Well-Being; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephonic CBT (Active Comparator): Computer guided, cognitive behavioral therapy (CBT) delivered by a clinician-administered telephone intervention.
  Interventions: Behavioral: Telephonic CBT
- Wait List Control (Sham Comparator): Randomized wait list control with measurement of study outcomes at week 0, 3 and 5 after the initiation of waiting.
  Interventions: Behavioral: Wait List Control

INTERVENTIONS:
Behavioral: Telephonic CBT — Cognitive behavioral therapy, guided by computer, using the TAD protocol for treatment of Adolescent Depression, modified for delivery by a nurse or master's level clinician over the telephone in 15-18 sessions lasting 30-45 minutes at weekly intervals. Includes regular and standardized weekly monitoring by the treating clinician of depressive symptoms and factors affecting suicide risk.
  Other Names: iTAD; ITEMS-TAD; Computer-guided CBT; TAD
  Arms: Telephonic CBT
Behavioral: Wait List Control — Wait list control with measurement of key outcomes at baseline (week 0), and then weeks 3 and 5.
  Arms: Wait List Control

SUMMARY:
The purpose of this study is to evaluate a computer-guided, telephone-based therapy for adolescent depression, delivered in a pediatric primary setting in the community.

DETAILED DESCRIPTION:
This Phase II SBIR project represents the continuing development of an Information Technology Enabled Disease Management System for Treatment of Adolescent Depression (iTAD) following a highly successful Phase I award in which all Specific Aims were met. The need for this system innovation arises from the substantial costs that inadequately treated adolescent Major Depressive Disorder (MDD) has on the course of adolescent development and society as a whole. Effective treatments involving the combined use of a Selective Serotonin Reuptake Inhibitor (SSRI) and the administration of Cognitive Behavioral Therapy (CBT) is considered the "modal treatment" for adolescent MM. Yet, multiple barriers interfere with the implementation and dissemination of this "gold standard' of care. These barriers include: under recognition of depressive symptoms by parents and pediatricians, inability to assess adolescent depression accurately and reliably in primary care settings, safety concerns related to pharmacologic treatment, monitoring of symptom changes and adverse treatment effects, such as irritability and suicidal behavior, treatment non-compliance, lack of access to an integrated medical and treatment history; and an alarming shortage of properly trained child and adolescent psychiatrists capable of implementing optimal treatment safely, reliably, and effectively.

In this current project, the investigators are making tailored forms of CBT broadly and easily accessible to the community, using the iTAD (previously "ITEMS-TAD") which is intended to address these problems. Development of the system has continued and we have modified the existing prototype that was created with funding from federal sources (Phase 1). The technological infrastructure of the prototype includes a Computer Assisted Telephone Interview (CATI) platform, a database consisting of patients' real time medical and treatment history, and an underlying set of intelligent algorithms that tailors the intensity of the treatment resources and approaches administered in individual cases, with a special focus on identifying those enrolled adolescents needing more intensive or urgent care. When interacting with patients over the telephone, primary care nurses use the CATI to facilitate the reliable assessment of patient status and administer manualized, empirically informed interventions. The programming for the platform that delivers this intervention is complete and the debugging and refinement underway. The content for the remaining iTAD program has been developed and is being programmed. A Rapid Iterative Evaluation & Testing (RITE) study was undertaken to refine the content of the application and assess the usability of the technology involved in its delivery; A field trial is underway to evaluate empirically indicators of efficacy and patient acceptance related to the ITEMS-TAD approach. The clinical trial of iTAD will begin in early April 2012. The investigators are currently enrolling depressed adolescents who will begin the trial shortly.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder
* Age 12-17 years, inclusive, at time of first study visit
* Ability to receive care as an outpatient
* Ability to participate in at least 1 session by phone per week for approximately 12 weeks
* Ability to participate in at least 1 session by phone per week for approximately 12-16 weeks
* Ability to speak English fluently and to provide written and/or verbal feedback on the instrument and the process.
* Pediatrician impression of normal IQ for developmental level

Exclusion Criteria:

* Current or past diagnosis of: bipolar disorder, severe conduct disorder, pervasive developmental disorders, of thought disorder
* Current treatment with Cognitive Behavioral Therapy (CBT)
* Confounding medical condition (such as pregnancy, Lyme disease, etc.)
* Non-English speaking patient or parent/guardian
* No access to phones
* Dangerousness to self or others if they have been hospitalized for dangerousness within three months of consent
* Deemed to be "high risk" because of a suicide attempt requiring medical attention within 6 months of consent or clear intent or an active plan to commit suicide
* History of self-harm, suicidal attempts, or suicidal ideation
* Specialty care for substance abuse (i.e. without participation of primary care providers)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in measures of depression over the course of treatment among teens with Major Depressive Disorder. | 12 weeks
  The measure used is the PHQ-9 (Kroenke, et al.), a standard and validated measure for use in screening for or monitoring adolescent depression. Teens that score positively on Item #9 (a self-harm risk item), will be further evaluated by the clinician using two interactive and validated methods for standardized assessment of suicide risk: a brief version of the Beck Hopelessness scale and the C-CASA (Columbia University). Teens needing referral to a behavioral health specialist will be referred by the nurse and/or the pediatrician for further evaluation and treatment.

SECONDARY OUTCOMES:
Evidence of program efficacy as indicate by changes in subjects' knowledge of depression. | 12 weeks
  A Depression Knowledge Test (DKT) will be used to assess changes in the level of knowledge teens have about depression and its treatment. The DKT consists of 10 open response questions based on materials from the TADS Adolescent Workbook. Sample questions include "We know there are four main causes of depression. List as many as you can," and "There are some learned patterns that people need to change to overcome depression. List as many patterns as you can."
Evidence of program efficacy as indicated by development of self-efficacy skills. | 12 weeks
  A Skill Self-Efficacy Questionnaire (SSEQ) will be used to assess changes in the level of self-confidence teens have in their ability to use the cognitive behavioral skills taught in the demo program. Using the same assessment schedule as the DKT, teens will be asked to rate self-confidence in their ability to "set goals," "achieve goals," "know what they are feeling," "know how intensely they feel something," and "know what causes their feelings."
Evidence of program efficacy as indicated by the establishment of therapeutic alliance. | 12weeks
  Therapeutic alliance between adolescents and nurse managers will be measured by the Therapeutic Alliance Scale for Adolescents (TASA; Shrink et al., 2008. The TASA is explicitly designed to measure the strength of the therapeutic alliance among teens participating in CBT treatments. A maximum score is 6.0 based on a Likert scale from one to six. The list of items for this measure of therapeutic alliance indicates very high bonding between counselors and patients.
Evidence of program efficacy as indicated by fidelity and treatment quality. | 12 weeks
  The Cognitive Therapy Scale (CTR) will be used as a measure of treatment quality and fidelity of the calls by and interactions of the study nurses with the teens. The CTR has been considered a standard measure of competence in cognitive therapy for more than 20 years,(Young JE 1980; Dobson, Shaw et al. 1985; Vallis, Shaw et al. 1986). Recorded sessions will be rated on the scale by certified raters from the American Academy of Cognitive Therapy (ACT).
Evidence of program efficacy as indicated by program acceptance. | 12 weeks
  An acceptance questionnaire will be administered to teens to determine their overall perception and acceptance of the program. The questionnaire contains 9 questions, asking the subject to rate the usefulness of the program; comment on its quality, and suggest areas for improvement. The acceptance questionnaire uses a 7-point Likert scale for rating purposes ranging from (1 = not at all to 7 = extremely). It also includes three open-ended questions to capture what teens like the best or the least about the program, and their suggestions for improving the program.

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Locke, MD, Principal Investigator — iHope Network, Inc.; Thomas J. McLaughlin, ScD, Principal Investigator — iHope Network, Inc.
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Woburn Pediatric Associates, Woburn, Massachusetts